CLINICAL TRIAL: NCT07215156
Title: Comparative Study Between Metformin and Chlorhexidine Gel as Adjunctive to Conventional Non-Surgical Treatment of Stage II Grade B Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Metformin Versus Chlorhexidine Gel as Adjuncts to Scaling and Root Planing in Stage II Grade B Periodontitis
Acronym: MET-CHX Perio
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Duaa Luwai Osman Hashim, (B.D.S. 2011 ) NATIONAL RIBAT UNIVERSITY, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-564
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Stage II, Grade B Periodontitis; Chronic Periodontitis
Keywords: Periodontitis; Stage II Grade B Periodontitis; Chronic Periodontitis; Scaling and Root Planing (SRP); Non-surgical Periodontal Therapy; Metformin Gel; Chlorhexidine Gel; Local Drug Delivery; Periodontal Regeneration; Inflammatory Markers (MMP-8)
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Root Planing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1:1 ratio to one of three parallel groups: SRP alone, SRP + Metformin gel, or SRP + Chlorhexidine gel.
Who Masked: Participant
Masking Description: Single-blind design: participants are blinded to intervention allocation; clinicians applying treatment are aware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Control: Scaling and Root Planing (SRP) Only (Active Comparator): Participants receive conventional subgingival scaling and root planing (SRP) alone using hand and ultrasonic instruments, plus standardized oral hygiene instruction. No adjunctive local drug or gel is applied.
  Interventions: Procedure: Arm 1 Scaling and Root Planing (SRP)
- Arm 2 - Experimental: SRP + 1% Metformin Gel (Experimental): Participants receive conventional SRP followed by subgingival application of 1% metformin gel into selected periodontal pockets; a periodontal dressing is placed for one week. Participants receive standardized oral hygiene instruction.
  Interventions: Drug: Arm 2 Metformin Gel 1% (locally delivered)
- Arm 3 - Experimental: SRP + 0.2% Chlorhexidine Gel (Experimental): Participants receive conventional SRP followed by subgingival application of 0.2% chlorhexidine gel into selected periodontal pockets; a periodontal dressing is placed for one week. Participants receive standardized oral hygiene instruction.
  Interventions: Drug: Arm 3 Chlorhexidine Gel 0.2% (locally delivered)

INTERVENTIONS:
Procedure: Arm 1 Scaling and Root Planing (SRP) — Full-mouth supragingival and subgingival debridement performed with ultrasonic and hand instruments (Gracey curettes). SRP performed to remove plaque and calculus and root-surface decontamination. Standardized oral hygiene instruction is provided after the procedure.
  Arms: Arm 1 - Control: Scaling and Root Planing (SRP) Only
Drug: Arm 2 Metformin Gel 1% (locally delivered) — 1% metformin hydrochloride formulated in a gellan-gum gel base (as per protocol). After SRP, gel is delivered subgingivally with a sterile syringe (23-gauge cannula) and left undisturbed for approximately 5 minutes; a periodontal dressing is placed for one week. Gingival crevicular fluid sampling and clinical follow-up at 1, 3, and 6 months.
  Arms: Arm 2 - Experimental: SRP + 1% Metformin Gel
Drug: Arm 3 Chlorhexidine Gel 0.2% (locally delivered) — 0.2% chlorhexidine digluconate gel prepared in carbopol base. After SRP, gel is delivered subgingivally with a sterile syringe and left undisturbed for approximately 5 minutes; a periodontal dressing is placed for one week. Clinical follow-up at 1, 3, and 6 months.
  Arms: Arm 3 - Experimental: SRP + 0.2% Chlorhexidine Gel

SUMMARY:
This clinical trial is designed to evaluate two locally delivered gels, metformin and chlorhexidine, as adjunctive therapies to scaling and root planing (SRP) in patients with Stage II, Grade B periodontitis. Periodontitis is a chronic inflammatory condition that damages the supporting tissues of the teeth. Although SRP is the standard non-surgical treatment, it may not fully eliminate harmful bacteria or prevent disease recurrence.

Chlorhexidine is a widely used antimicrobial gel, while metformin, a medication commonly prescribed for diabetes, has shown anti-inflammatory and bone-supportive effects when used locally in the gums. This study will directly compare the effectiveness of 1% metformin gel and 0.2% chlorhexidine gel, both applied subgingivally after SRP, against SRP alone.

Sixty adult participants diagnosed with Stage II, Grade B periodontitis will be randomly assigned into three groups: SRP only (control), SRP plus metformin gel, and SRP plus chlorhexidine gel. Clinical outcomes (plaque index, gingival index, probing pocket depth, and clinical attachment level), inflammatory markers (MMP-8 in gingival crevicular fluid), and radiographic bone density will be measured at baseline, 1 month, 3 months, and 6 months.

The goal is to determine whether metformin gel or chlorhexidine gel provides superior improvements in periodontal healing when compared with SRP alone. Findings from this trial may guide evidence-based decisions on optimizing non-surgical periodontal therapy.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-blind clinical trial conducted at the Department of Oral Medicine, Periodontology, Oral Diagnosis, and Oral Radiology, Faculty of Dentistry, Kafrelsheikh University, Egypt. Sixty participants aged 18-60 years with Stage II, Grade B periodontitis will be enrolled. Participants will be randomly allocated (1:1:1) into three groups:

Group A (Control): SRP only

Group B (Test 1): SRP + 1% Metformin Gel

Group C (Test 2): SRP + 0.2% Chlorhexidine Gel

Subgingival gels will be applied after SRP using sterile syringes, followed by periodontal pack placement for one week. All patients will receive standardized oral hygiene instructions.

Outcome Measures:

Primary Outcomes: Clinical attachment level (CAL) changes, reduction in inflammatory markers (MMP-8), and radiographic bone density gain.

Secondary Outcomes: Probing pocket depth (PPD), plaque index (PI), and gingival index (GI).

Follow-up assessments will be performed at 1, 3, and 6 months. Data will be statistically analyzed using ANOVA and paired t-tests, with significance at p < 0.05.

The trial has been reviewed and approved by the Scientific Research Ethics Committee, Faculty of Dentistry, Kafrelsheikh University (Approval No. KFSIRB200-564, dated 24 February 2025).

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-60 years.

Diagnosis of Stage II, Grade B periodontitis.

Probing pocket depths ≤ 5 mm with clinical attachment loss of 3-4 mm in selected sites.

Generally healthy individuals without systemic conditions affecting periodontal health.

Exclusion Criteria:

Current smokers or users of tobacco products.

Pregnant or lactating women.

Known allergy to metformin or chlorhexidine.

Use of antibiotics or anti-inflammatory drugs within the past 3 months.

History of periodontal therapy within the past 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gingival Crevicular Fluid MMP-8 Levels | Baseline, 1 month, and 3 months
  Active MMP-8 concentrations will be quantified in gingival crevicular fluid using ELISA. PerioPaper strips will be used for collection. Reduction in MMP-8 indicates decreased periodontal inflammation.
Change in Clinical Attachment Level (CAL) | Baseline, 1 month, 3 months, and 6 months
  CAL will be measured from the cementoenamel junction to the base of the periodontal pocket using a UNC-15 probe. Improvement in CAL reflects periodontal tissue healing and attachment gain.
Change in Alveolar Bone Density | Baseline, 3 months, and 6 months
  Standardized periapical digital radiographs will be analyzed using Digora software to calculate mean gray-level values in the region of interest (1 mm below CEJ, 7 mm apically). An increase indicates bone density improvement.

SECONDARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline, 1 month, 3 months, and 6 months
  Probing depth will be measured at six sites per tooth using a UNC-15 probe. Reduction in pocket depth indicates clinical improvement in periodontal status.
Change in Gingival Index (GI) Score | Baseline, 1 month, 3 months, and 6 months
  Gingival inflammation will be assessed using the Löe and Silness Gingival Index. Decreased GI score reflects reduction in gingival inflammation.
Change in Plaque Index (PI) Score | Baseline, 1 month, 3 months, and 6 months
  Oral hygiene status will be evaluated using the Silness and Löe Plaque Index. Reduction in PI indicates improved plaque control.

IPD SHARING:
Plan to Share IPD: No